CLINICAL TRIAL: NCT02783846
Title: The Effects of Different Dexmedetomidine on the Propofol Requirement for Loss of Consciousness Undergoing Bispectral Index
Brief Title: The Effects of Different Doses of Dexmedetomidine on Propofol Requirement for Loss of Consciousness Undergoing Bispectral Index: a Double-blinded, Placebo-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MHX00123
Record Dates: First submitted 2016-05-16; First posted 2016-05-26 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-08

CONDITIONS: Loss of Consciousness
Keywords: Propofol; Dexmedetomidine; Dose; Bispectral index monitor
MeSH Terms: conditions — Unconsciousness | interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group control (Placebo Comparator): 24 eligible patients are received equal volumes of saline intravenously for 10 minutes
  Interventions: Other: normal saline
- Group dexmedetomidine 0.5 µg/kg (Active Comparator): 24 eligible patients are received dexmedetomidine 0.5 µg/kg intravenously for 10 minutes
  Interventions: Drug: dexmedetomidine 0.5 µg/kg
- Group dexmedetomidine 1.0 µg/kg (Active Comparator): 25 eligible patients are received dexmedetomidine 1.0 µg/kg intravenously for 10 minutes
  Interventions: Drug: dexmedetomidine 1.0 µg/kg

INTERVENTIONS:
Other: normal saline — receive equal volume of normal saline
  Arms: Group control
Drug: dexmedetomidine 0.5 µg/kg — receive dexmedetomidine 0.5 µg/kg
  Arms: Group dexmedetomidine 0.5 µg/kg
Drug: dexmedetomidine 1.0 µg/kg — receive dexmedetomidine 1.0 µg/kg
  Arms: Group dexmedetomidine 1.0 µg/kg

SUMMARY:
The purpose of this study is to evaluate the effects of different dexmedetomidine on the propofol requirement for loss of consciousness undergoing bispectral index.

DETAILED DESCRIPTION:
It has been shown that dexmedetomidine was an efficacious and safe adjuvant in general anaesthesia. Administration of dexmedetomidine during the preoperative period has been demonstrated to reduce the requirement of opioid analgesics and other sedative and hypnotic drugs.Therefore, the study is designed to measure the effect of intravenous dexmedetomidine premedication on the propofol dose requirement and bispectral index at loss of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Aged 18-65 years
* Body Mass Index 18.0～24.5 kg/m2
* Without hearing impairment

Exclusion Criteria:

* Bradycardia
* Atrioventricular block
* Neurologic disorder and recent use of psychoactive medication
* Allergic to the drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The propofol requirement for pretreatment of dexmedetomidine by micro-pump until loss of consciousness | To infuse dexmedetomidine and saline completely ten minutes after

SECONDARY OUTCOMES:
The bispectral index values when patients loss of consciousness | To infuse dexmedetomidine and saline completely ten minutes after

IPD SHARING:
Plan to Share IPD: No
safety

REFERENCES:
- [Derived] Gu Y, Yang F, Zhang Y, Zheng J, Wang J, Li B, Ma T, Cui X, Lu K, Ma H. The effects of different doses of dexmedetomidine on the requirements for propofol for loss of consciousness in patients monitored via the bispectral index: a double-blind, placebo-controlled trial. BMC Anesthesiol. 2020 Apr 25;20(1):96. doi: 10.1186/s12871-020-01013-x. PMID 32334510